CLINICAL TRIAL: NCT01107522
Title: A Phase I Study of Oral Carboxyamidotriazole Orotate (CTO) Titrated as a Single Agent in Patients With Advanced or Metastatic Solid Tumors and Titrated in Combination Therapy With Temodar® for Patients With Glioblastoma and Other Recurrent Malignant Gliomas or in Combination With Temodar® and Radiation Therapy for Patients With Newly Diagnosed Glioblastoma and Malignant Gliomas
Brief Title: Safety and Tolerability of Carboxyamidotriazole Orotate (CTO) in Solid Tumors or With Temodar® in Glioblastoma or Other Recurrent Malignant Gliomas or in Combination With Temodar® and Radiation Therapy for Patients With Newly Diagnosed Glioblastoma and Malignant Gliomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tactical Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T09-10644
Record Dates: First submitted 2010-04-16; First posted 2010-04-21 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumors, Glioblastoma, Recurrent Malignant Gliomas
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Temozolomide; Radiotherapy

ARMS (3):
- Arm A (Experimental): Single Agent CTO
  Interventions: Drug: CTO
- Arm B (Experimental): Combination CTO and Temodar®
  Interventions: Drug: CTO and Temodar®
- Arm C (Experimental): Combination CTO, Temodar®, Radiation therapy
  Interventions: Drug: CTO, Temodar®, Radiation therapy

INTERVENTIONS:
Drug: CTO — Oral administration daily for 28 day cycles; starting dose of CTO = 50 mg/m2
  Arms: Arm A
Drug: CTO and Temodar® — Oral administration of CTO daily for 28 day cycles, starting dose of CTO = 219 mg/m2.
  Temodar® administered orally at fixed dose of 150 mg/m2 daily for Days 1-5 in a 28 day cycle.
  Expansion Cohort of 6 patients on fixed dose of 600mg CTO/day Temodar® administered orally at fixed dose of 150 mg/m2 daily for Days 1-5 in a 28 day cycle
  Arms: Arm B
Drug: CTO, Temodar®, Radiation therapy — Oral administration of CTO daily for 28 day cycles; starting dose of CTO = 219 mg/m2 Temodar® administered orally at a dose of 75 mg/m2 daily during radiation therapy, then at 150mg/m2 for Days 1-5 of Cycle 1, and then up to 200 mg/m2 Days 1-5 of subsequent cycles Radiation: 3-dimensional conformal radiation therapy or, Radiation: intensity-modulated radiation therapy
  Arms: Arm C

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and the maximum tolerated dose/recommended phase II dose of carboxyamidotriazole orotate (CTO) as a single agent in patients with advanced or metastatic solid tumors; in combination with oral Temodar® in patients with glioblastoma or other recurrent malignant gliomas; or in combination with oral Temodar® and radiation therapy in patients with newly diagnosed glioblastoma or other malignant gliomas.

ELIGIBILITY:
Inclusion Criteria (Treatment Arm A)

1. Patients must have histologically-confirmed solid tumors that are advanced or metastatic, and refractory after standard therapy, or for which there is no standard therapy.
2. Patients must have measurable disease as defined by RECIST version 1.1.
3. Patients must have received prior anticancer therapy or not be eligible for any established conventional therapy whether surgical or pharmacologic.
4. Patients must have recovered from all acute adverse effects (excluding alopecia) of prior therapies to baseline or <=grade 1 prior to study entry.
5. Patients must have a performance status of 0, 1, or 2.
6. Patients must be men and women >=18 years of age.
7. Patients must have adequate bone marrow function, defined as an absolute neutrophil count >=1.5 x 10^9/L and a platelet count >= 100 x 10^9/L.
8. Patients must have adequate renal function, defined as serum creatinine <= 1.2 mg/dL (if > 1.2 mg/dL, a calculated creatinine clearance [by the Cockcroft-Gault method] must be >=60 mL/min/1.73 m^2).
9. Patients must have adequate hepatic function, defined as plasma total bilirubin <=1.5 mg, alanine transaminase (ALT) and aspartate transaminase (AST) <=2.5 X ULN. Patients with Gilbert's disease outside these limits are judged to be ineligible.
10. Female patients of childbearing potential must have a negative serum or urine pregnancy test result at time of pre-treatment screening.
11. Patients with reproductive potential must agree to use at least one form of barrier contraception prior to study entry and for up to 30 days beyond the last administration of study drug.
12. Patients must be judged to be capable by the Investigator of providing informed consent and must be willing to provide written informed consent prior to the start of any study specific procedures.
13. Patients should have a life expectancy of at least 12 weeks.

Exclusion Criteria (Treatment Arm A)

1. Patients may not have had prior chemotherapy, hormonal therapy, radiation therapy, or biologic therapy in the 4 weeks prior to study entry with the exception of mitomycin C or nitrosoureas, for which patients must be 6 weeks from prior treatment. For patients who have been treated with targeted therapy, 5 half-lives of that therapy (or 28 days, whichever is shorter) must have passed prior to enrollment in the study.
2. Patients may not have any concomitant condition that could compromise the objectives of this study and the patients' compliance and ability to tolerate this therapy and complete at least 2 cycles of therapy, including, but not limited to the following:

   * Congestive heart failure or uncontrolled angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension, or dysrhythmias.
   * Active infection.
   * Unstable diabetes mellitus
   * Psychiatric disorder that may interfere with consent and/or protocol compliance.
3. Pregnant or breastfeeding women.
4. Patients with another malignancy in the past 3 years except: curatively treated non-melanoma skin cancer; or carcinoma in situ, of either cervix or breast, that does not require further treatment.
5. Patients with known HIV, HBV, or HCV infection.
6. Patients with an underlying diagnosis or disease state associated with an increased risk of bleeding.
7. Patients with central nervous system metastases. Baseline CT or MRI scan of brain is required only in the case of clinical suspicion of central nervous system metastases. Patients with evidence of brain involvement, leptomeningeal disease, or seizure disorder are also excluded.
8. Patients may not be treated with known CYP3A4 inhibitors or inducers.

Inclusion and Exclusion Criteria for Combination CTO Plus Temodar® (Treatment Arm B): Inclusion Criteria (Treatment Arm B)

In addition to the inclusion criteria for adequate organ function as defined for the patients with advanced or metastatic solid tumors, patients enrolled in Arm B (Combination Therapy CTO Plus Temodar-R) must meet the following inclusion criteria:

1. Patients must have histologically proven malignant glioblastoma or other recurrent malignant gliomas.
2. Measurable tumor must be present on gadolinium-enhanced MRI.
3. Patients must have a life expectancy of at least 8 weeks.
4. Patients must have a Performance Status of 0, 1, or 2 (ECOG scale).
5. Patients must be men and women >=18 years of age.
6. Patients must have recovered from all acute adverse effects (excluding alopecia) of prior therapies to baseline or <=grade 1 prior to study entry.
7. Patients must have shown unequivocal radiographic evidence for tumor progression by MRI scan to be performed within 14 days prior to registration and must be on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI scan is required.
8. Patients who have undergone recent resection for recurrent or progressive malignant tumor will be eligible as long as all of the following conditions apply:

   1. They have recovered from the effects of surgery
   2. The extent of residual disease is assessed post-operatively, with an MRI scan done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated.
9. Patients must have had prior radiation therapy with or without chemotherapy and must have progressed following radiation therapy and must have an interval of >=12 weeks from the completion of radiation therapy to registration date to minimize the possibility of pseudo-progression.
10. Patients under treatment with anti-epileptic drugs which are not known CYP3A4 inhibitors or inducers must have been receiving a stable dose for at least 2 weeks with no evidence of seizures at the time of registration.

Exclusion Criteria (Treatment Arm B)

1. Patients may not have had prior chemotherapy, hormonal therapy, or biologic therapy in the 4 weeks prior to study entry with the exception of mitomycin C or nitrosoureas, for which patients must be 6 weeks from prior treatment. For patients who have been treated with targeted therapy, 5 half-lives of that therapy (or 28 days, whichever is shorter) must have passed prior to enrollment in the study. Additional exceptions: The following specific drugs are permitted shorter recovery times: 14 days for vincristine, 21 days for procarbazine, and 7 days for non-cytotoxic agents such as interferon, tamoxifen, thalidomide, and cis-retinoic acid.
2. Patients may not have any concomitant condition that could compromise the objectives of this study and the patients' compliance and ability to tolerate this therapy and complete at least 2 cycles of therapy, including, but not limited to the following:

   * Congestive heart failure or uncontrolled angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension, or dysrhythmias.
   * Active infection.
   * Unstable diabetes mellitus.
   * Psychiatric disorder that may interfere with consent and/or protocol compliance.
3. Pregnant or breastfeeding women.
4. Patients with another malignancy in the past 3 years except: curatively treated non-melanoma skin cancer; or carcinoma in situ, of either cervix or breast, that does not require further treatment.
5. Patients with known HIV, HBV, or HCV infection.
6. Patients with an underlying diagnosis or disease state associated with an increased risk of bleeding.
7. Uncontrolled seizure activity.
8. Patients may not be treated with known CYP3A4 inhibitors or inducers.

Inclusion and Exclusion Criteria for Combination CTO and Temodar® in combination with radiation therapy (Treatment Arm C):

Inclusion Criteria (Treatment Arm C)

In addition to the inclusion criteria for adequate organ function as defined for the patients with advanced or metastatic solid tumors, patients enrolled in Arm C (Combination Therapy CTO and Temodar® in combination with radiation therapy) must meet the following inclusion criteria:

1. Patients must have histologically proven newly diagnosed glioblastoma or other malignant gliomas. Note: Patients with anaplastic oligodendroglioma with 1p/19q deletion or unknown 1p/19q status are not eligible
2. Patients must have a life expectancy of at least 8 weeks
3. Patients must have a Performance Status of 0, 1, or 2 (ECOG scale).
4. Patients must be men and women >=18 years of age.
5. Patients must have undergone an MRI scan performed within 14 days prior to registration and must be on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required.
6. Patients under treatment with anti-epileptic drugs which are not known CYP3A4 inhibitors or inducers must have been receiving a stable dose for at least 2 weeks with no evidence of seizures at the time of registration.

Exclusion Criteria (Treatment Arm C)

1. Patients may not have had any prior chemotherapy, hormonal therapy, or biologic therapy for gliomas.
2. Patients may not have any concomitant condition that could compromise the objectives of this study and the patients' compliance and ability to tolerate this therapy and complete at least 2 cycles of therapy, including, but not limited to the following:

   * Congestive heart failure or uncontrolled angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension, or dysrhythmias.
   * Active infection.
   * Unstable diabetes mellitus.
   * Psychiatric disorder that may interfere with consent and/or protocol compliance.
3. Pregnant or breastfeeding women.
4. Patients with another malignancy in the past 3 years except: curatively treated non-melanoma skin cancer; or carcinoma in situ, of either cervix or breast, that does not require further treatment.
5. Patients with known HIV, HBV, or HCV infection.
6. Patients with an underlying diagnosis or disease state associated with an increased risk of bleeding.
7. Uncontrolled seizure activity.
8. Patients may not be treated with known CYP3A4 inhibitors or inducers.
9. Patients with anaplastic oligodendroglioma with 1p/19q deletion or unknown 1p/19q status are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD/RD of single agent CTO in patients with advanced or metastatic solid tumors; or CTO in combination with Temodar® in patients with glioblastoma or other recurrent malignant gliomas | Duration of the study
  To determine the highest tolerated dose of CTO, based on safety data and occurence of dose-limiting toxicity, in patients with advanced or metastatic solid tumors. In the second stage of the study, to determine the highest tolerated dose of CTO in combination with Temodar®, based on safety data and toxicity profile, in patients with glioblastoma or other recurrent malignant gliomas. In the third stage of the study, to determine the highest tolerated dose of CTO in combination with Temodar® and radiation therapy based on safety data and toxicity profile, in patients with newly diagnosed glioblastoma or other malignant gliomas.

SECONDARY OUTCOMES:
Preliminary tumor response | after every 2 cycles
  RECIST 1.1 (Arm A); Macdonald Criteria (Arms B and C)
Pharmacokinetics (maximum concentration, Tmax, AUC, T1/2, clearance, volume of distribution) | pre- and post-dose during cycle 1
  Plasma concentrations and PK parameters will be determined for single agent CTO (Arm A), or CTO in combination with Temodar® (Arm B); plasma concentrations and PK parameters will be determined for Temodar®, or CTO and Temodar® in combination with radiation therapy (Arm C).
Voluntary Exploratory objective | collected prior to enrollment
  To investigate effect of CTO on tumor growth based on genotype
Exploratory Objective | Duration of study
  To investigate effect of CTO alone and in combination with Temodar® on gene expression in scalp hair

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Taylor, MD, Principal Investigator — Oregon Health and Sciences University; Elena Pentsova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Walter Urba, MD, PhD, Principal Investigator — Providence Health & Services; Katharine McNeill, MD, Principal Investigator — NYU MEDICAL CENTER; Lisa DeAngelis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Timothy Chan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - New York University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Providence Cancer Center, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon

REFERENCES:
- [Derived] Omuro A, Beal K, McNeill K, Young RJ, Thomas A, Lin X, Terziev R, Kaley TJ, DeAngelis LM, Daras M, Gavrilovic IT, Mellinghoff I, Diamond EL, McKeown A, Manne M, Caterfino A, Patel K, Bavisotto L, Gorman G, Lamson M, Gutin P, Tabar V, Chakravarty D, Chan TA, Brennan CW, Garrett-Mayer E, Karmali RA, Pentsova E. Multicenter Phase IB Trial of Carboxyamidotriazole Orotate and Temozolomide for Recurrent and Newly Diagnosed Glioblastoma and Other Anaplastic Gliomas. J Clin Oncol. 2018 Jun 10;36(17):1702-1709. doi: 10.1200/JCO.2017.76.9992. Epub 2018 Apr 23. PMID 29683790